CLINICAL TRIAL: NCT02686346
Title: Phase I/II Feasibility Study of Brentuximab Vedotin in Refractory / Relapsed Hodgkin Lymphoma Patients Who Are Treated by Chemotherapy (ICE) in Second Line and Eligible for Autologous Transplantation
Brief Title: Brentuximab Vedotin in Refractory/Relapsed Hodgkin Lymphoma Treated by ICE
Acronym: BV-ICE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV-ICE
Record Dates: First submitted 2016-02-09; First posted 2016-02-19 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Hodgkin Disease
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Brentuximab Vedotin; Etoposide; Carboplatin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BV-ICE (Experimental): Phase I:
  4 cycles of treatment, every 21 days: Brentuximab Vedotin (BV) + Etoposide- Carboplatine - Ifosfamide (ICE) = BV-ICE for cycles 1 to 3 and BV alone at cycle 4;
  Phase II:
  4 cycles of treatment, every 21 days: BV-ICE for cycles 1 to 3, BV alone at cycle 4
  Interventions: Drug: Brentuximab Vedotin; Drug: Etoposide; Drug: Carboplatine; Drug: Ifosfamide

INTERVENTIONS:
Drug: Brentuximab Vedotin — Phase I:
  Cohort K: BV on Day 1: 1.2 mg/kg (cycle 1-3) and 1.8 mg/kg (cycle 4) Cohort K+1: BV on Day 1: 1.8 mg/kg (cycle 1-3) and 1.8 mg/kg (cycle 4) Cohort K-1: BV on Day 1: 0.8 mg/kg (cycle 1-3) and 1.8 mg/kg (cycle 4)
  Phase II:
  BV on Day 1: at the Maximal Tolerated Dose (MTD) defined at Phase I
  Other Names: BV; SGN35
Drug: Etoposide — 100 mg/m² Days 1-2-3 of Cycles 1-2-3
Drug: Carboplatine — max 800mg Day 2 of Cycles 1-2-3
Drug: Ifosfamide — 5 g/m² Day 2 of Cycles 1-2-3

SUMMARY:
This study is designed as a phase Ib/II trial. The first part (phase Ib) is a dose escalation design to explore the safety and assess the recommended phase 2 dose of Brentuximab Vedotin in Hodgkin lymphoma patients treated with ICE regimen.

The second part, depending on the selected dose after the completion of phase Ib part of the study, will further explore safety in addition to efficacy of the recommended dose of Brentuximab Vedotin in a selected population of patients treated with ICE with Hodgkin lymphoma.

DETAILED DESCRIPTION:
PHASE I:

3 cycles of Brentuximab Vedotin ICE every 3 weeks and one cycle of Brentuximab Vedotin alone at the doses described below.

Cohorts of between three and six evaluable patients will be recruited at each dose level.

Dose escalation rules:

Treat 3 patients at level K

1. If 0 patients experience dose-limiting toxicity (DLT), escalate to dose K+1
2. If 2 or more patients experience DLT, de-escalate to level K-1
3. If 1 patient experiences DLT, treat 3 more patients at dose level K A. If 1 of 6 experiences DLT, escalate to dose level K+1 B. If 2 or more of 6 experiences DLT, de-escalate to level K-1 Dose escalation will begin at level K.

Level K:

Brentuximab Vedotin: 1.2 mg/kg (cycle 1-3), 1.8 mg/kg (cycle 4) ICE (cycle 1-3): Etoposide 100 mg/m² (day1 to 3); Carboplatine max 800mg (day 2); Ifosfamide + Mesna 5 g/m² (day 2)

Level K -1:

Brentuximab Vedotin: 0.8 mg/kg (cycle 1-3), 1.8 mg/kg (cycle 4) ICE (cycle 1-3): Etoposide 100 mg/m² (day1 to 3); Carboplatine max 800mg (day 2); Ifosfamide + Mesna 5 g/m² (day 2)

Level K +1:

Brentuximab Vedotin: 1.8 mg/kg (cycle 1-3), 1.8 mg/kg (cycle 4) ICE (cycle 1-3): Etoposide 100 mg/m² (day1 to 3); Carboplatine max 800mg (day 2); Ifosfamide + Mesna 5 g/m² (day 2)

Dose finding rule:

Provisional dose levels are listed in previous tables. Dose-escalation will continue until Maximal Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) is reached or the full doses of BV and ICE are delivered without DLT

PHASE II:

3 cycles of Brentuximab Vedotin + ICE every 3 weeks and one cycle Brentuximab Vedotin alone.

The recommended dose of BV and ICE will be determined by the phase I Brentuximab Vedotin: MTD mg/kg (cycle 1-3), 1.8 mg/kg (cycle 4) ICE (cycle 1-3): Etoposide 100 mg/m² (day1 to 3); Carboplatine max 800mg (day 2); Ifosfamide + Mesna 5 g/m² (day 2) The recommended dose of BV and ICE will be determined by the phase I.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cluster of differentiation antigen 30 + (CD30+) HL, primarily refractory to first line chemotherapy or in first relapse after any polychemotherapy regimen
* Measurable disease defined as at least one single node or tumor lesion on CT scan > 1.5 cm
* Fluorodeoxyglucose (FDG)-PET/ CT realized at relapse and positive.
* Age ≥ 18 years and up to 65 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2 (see appendix 19.5)
* Life expectancy of > 3 months with treatment
* No major organ dysfunction, unless HL-related
* Normal cardiac and pulmonary function for auto transplantation
* Total bilirubin < 1.5 x ULN (unless due to lymphoma involvement of the liver or a known history of Gilbert's syndrome)
* Alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2 x ULN (unless due to lymphoma involvement of the liver : ≤ 5 x ULN)
* Creatinine clearance > 60 mL/min
* Absolute neutrophil count ≥ 1.5x109/L, unless caused by diffuse bone marrow infiltration by the HL
* Platelets ≥ 100x109/L, unless caused by diffuse bone marrow infiltration by the HL
* Hemoglobin must be ≥ 8g/dL
* Written informed consent
* Able to adhere to the study visit schedule and other protocol requirements
* Eligible for high dose chemotherapy and autologous peripheral blood stem cell transplantation
* Resolution of toxicities from first-line therapy
* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
* Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Peripheral sensory or motor neuropathy grade ≥ 2
* Any chemotherapy, radiotherapy, immunotherapy or investigational, therapy for treatment of lymphoma within 28 days prior Cycle1 Day1
* Patient who have been treated by first line of treatment with brentuximab vedotin alone or in combination
* Female patients who are both lactating and breast feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test 4 days prior the start of study drug
* Patients with active, uncontrolled infections (requiring systemic antibiotics within two weeks prior to treatment)
* Prior history of another cancer unless the subject has been free of the disease for ≥ 3 years (with the exception of non-melanoma skin cancer, completely resected melanoma TNMpT1 or carcinoma in situ of the uterine cervix)
* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of Progressive multifocal leukoencephalopathy
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
* Known history of human immunodeficiency virus (HIV), or known active Hepatitis C Virus, or active Hepatitis B Virus (HBV) infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
* Patients with a psychiatric disorder that would preclude compliance with drug delivery
* Patients who have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study such as:

  1. unstable angina pectoris, symptomatic congestive heart failure (NYHA II, III, IV), myocardial infarction ≤ 2 years prior to first study drug administration, serious uncontrolled cardiac arrhythmia, angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  2. cerebrovascular accident ≤ 6 months before study drug start recent evidence (within 6 months before first dose of study drug)
  3. a left-ventricular ejection fraction <50%
  4. severely impaired pulmonary function as defined as spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) that is 50% or less of the normal predicted value and/or O2 saturation that is 90% or less at rest on room air
  5. any active (acute or chronic) or uncontrolled disorders that impair the ability to evaluate the patient or for the patient to complete the study
  6. any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
  7. nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by this study drug, such as severe hypertension that is not controlled with medical management and thyroid abnormalities when thyroid function cannot be maintained in the normal range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Phase I : Maximal Tolerated Dose (MTD) determination | 4 months
  To determine the MTD and/or Recommended Phase II dose (RP2D dose) of BV when administered to adult patients treated with ICE in refractory or relapsed Hodgkin's lymphomas.
Phase II = fraction of responding patients according to Lugano classification (metabolic Complete Response) | 2 months
  To evaluate the efficacy of BV in patient treated with ICE as first salvage treatment (establish the fraction of responding patients - metabolic Complete Response (CR)) as judged by the center by Lugano classification after the second cycle

SECONDARY OUTCOMES:
Phase I : Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 4 months
  To characterize the safety and tolerability of BV in patient treated with ICE.
Phase I = Preliminary Overall Response Rate (ORR) | 4 months
  To assess preliminary anti-tumor activity of BV in patient treated with ICE.
Phase II = ORR | 4 months
  To assess the ORR (Complete Response and Partial Response) after 3 cycles of BV and ICE and one cycle of BV
Phase II : Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 4 months
  To assess the toxicity profile of BV in patient treated with ICE
Phase II = number of patients with hematological recovery after each cycle | 4 months
  To assess hematological recovery after each cycle of BV and ICE
Phase II = Feasibility of Autologous Stem Cell Transplant (ASCT) after BV-ICE = fraction of patients for whom harvest is possible | 4 months
  To assess the feasibility of harvesting an autologous peripheral blood stem cell graft after BV in patient treated with ICE
Phase II = Fraction of patients eligible for ASCT | 4 months
  To assess the fraction of patients (Complete Response/Partial Response) eligible for ASCT who actually underwent one or two ASCT
Phase II = Number of patients Positron Emission Tomography (PET) 4- after PET 2+ | 4 months
  To assess the number of patients with PET 4 negative if the PET 2 is positive
Phase II = Progression Free Survival (PFS) | 2 years
  Number of participants who did not progressed after 2 years
Phase II = Overall Survival (OS) | 2 years
  Number of participants alive after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Brice, MD, Principal Investigator — Lymphoma Study Association; Aspasia Stamatoullas Bastard, MD, Principal Investigator — Lymphoma Study Association
Locations (19):
- Belgium (2):
  - Clinique Universitaire Saint-Luc, Brussels
  - CHU Dinant Godinne, Yvoir
- France (17):
  - Institut d'Hématologie de Basse Normandie - CHU Côte de Nacre, Caen
  - APHP-Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - CHU Saint Eloi, Montpellier
  - CHU De Nantes, Nantes
  - Hôpital Necker, Paris
  - APHP - Hôpital Saint Louis, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de La Milétrie, Poitiers
  - CHU De Rennes, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU De Strasbourg, Strasbourg
  - IUCT Toulouse, Toulouse
  - CHU De Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stamatoullas A, Ghesquieres H, Feugier P, Andre M, Le Bras F, Gac AC, Borel C, Gastinne T, Quittet P, Morschhauser F, Ribrag V, Guidez S, Nicolas-Virelizier E, Berriolo-Riedinger A, Vander Borght T, Edeline V, Brice P. Final results of brentuximab vedotin combined with ifosfamide-carboplatin-etoposide in first refractory/relapsed Hodgkin lymphoma: a lymphoma study association phase I/II study. Leuk Lymphoma. 2022 Dec;63(13):3063-3071. doi: 10.1080/10428194.2022.2107204. Epub 2022 Aug 17. PMID 35975738